CLINICAL TRIAL: NCT03360968
Title: Heartrate Variability During Conventional and Variable Pressure Support Mechanical Ventilation: a Cross-over Study
Brief Title: Heartrate Variability During Conventional and Variable Pressure Support Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Vienna University of Technology (Other)
Responsible Party: Principal Investigator, Maximilian Schnetzinger BSc, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EK Nr: 1827/2017
Record Dates: First submitted 2017-11-22; First posted 2017-12-04 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A-B (Experimental): Patient is treated with 1 hour SPN-CPAP/PS followed by 1 hour of Variable-PS ventilation mode
  Interventions: Procedure: Variable-PS; Procedure: SPN-CPAP/PS
- Treatment B-A (Experimental): Patient is treated with 1 hour Variable-PS followed by 1 hour of SPN-CPAP/PS ventilation mode
  Interventions: Procedure: SPN-CPAP/PS; Procedure: Variable-PS

INTERVENTIONS:
Procedure: Variable-PS — Variable-PS mode switched on for 1 hour
  Arms: Treatment A-B
Procedure: SPN-CPAP/PS — SPN-CPAP/PS mode switched on for 1 hour
Procedure: Variable-PS — Variable-PS mode switched on for 1 hour
  Arms: Treatment B-A

SUMMARY:
Rationale Studies show that about a third of all postoperative complications are due to cardiovascular reasons. Furthermore it was shown that more than 50% of postoperative deaths are associated with severe cardiovascular incidents. After surgical interventions seriously ill patients are transferred to intensive care units and mechanically ventilated. However there is not much evidence about the impact of mechanical ventilation on the cardiovascular system and cardiovascular complications. Artificial mechanical ventilation greatly differs from physiological breathing. In contrast to physiological negative pressure ventilation of th lung, mechanical positive pressure ventilation can cause ventilator induced lung injuries. Furthermore a significant deterioration of lung-heart-interaction during mechanical ventilation is known.

Relevance Mechanical ventilation leads to a decreased heartrate-variability, which has to be understood as increased stress on the cardiovascular system. Recently, a new ventilation mode called "variable pressure support ventilation" (VPSV) also known as "noisy pressure support ventilation". This new ventilation mode is similar to the ventilator mode "spontaneous-continuous positive airway pressure/pressure support" (SPN-CPAP), which is often used in a intensive care unit routine. Though VPSV differs through varying applicated pressure support and therefore tidal volumes. Therefore the new ventilation mode rather imitates physiological situation, since tidal volumes vary in physiological breathing, which has positive impact on heart-lung-interaction.

DETAILED DESCRIPTION:
Spontaneous-continuous positive airway pressure support (SPN-CPAP/PS) is the routine ventilator mode used in critically ill patients submitted to an intensive care unit (ICU). It guarantees a positive end expiratory pressure, which prevents atelectasis and minimizes weaning time, by supporting the patient's respiratory drive.

A few years ago, this very established ventilation technique was modified by simply altering the rhythm and volume of gas application: instead of administering same tidal volumes in equal time intervals a variation of applied volume as well as altering frequency in ventilation is introduced. This ventilation method is termed noisy pressure support ventilation (noisy PSV) or variable pressure support ventilation (variable PSV). The variation of pressure support will be within a range around a mean support-pressure (Psupp) and won't exceed a maximum pressure (Pmax), which are both adjusted before starting noisy PSV.

Any variation of breathing is physiological and may occur during speaking, moving and many other factors. As novel concept, the investigator proposes that such variation of ventilation rhythm and volume may have an important impact on heart rate variability (HRV), which is known as to be an indicator of a healthy heart. Since it has been observed that HRV is an important predictor of mortality in coronary care units, investigation of HRV became more important. Recently it was found that low HRV is associated with an increasing mortality and proposed low HRV to be a marker for critical illness.

The analysis and further investigation of HRV has therefore become an important issue in modern medicine. Mechanical ventilation plays a pivotal role in ICUs and should be further improved. Mechanical ventilation per se is stressful for the cardiovascular system. Cardiovascular homeostasis is of major importance and the investigator hypothesises that noisy PSV will decrease the stress applied to the human heart measured via heart rate variability.

In this interventional clinical study, the investigator will apply, in a randomized fashion, conventional PSV and variable PSV each for a duration of one hour. During ventilation the investigator will record all data of the patients monitor, including the electrocardiogram (ECG), which is routinely monitored in patients, and respiratory data, to determine HRV parameters retrospectively. All other ventilatory, hemodynamic and pharmacological treatment will be part of the clinical routine. As two modes of ventilation will be compared, this study is an interventional clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing therapy at an ICU; patients intubated and ventilated using SPN-CPAP/PS ventilator mode; patients with sinus rhythm in electrocardiogram

Exclusion Criteria:

* patients with active heart pace maker / defibrillator; patients with absent sinus rhythm in electrocardiogram; patients with known severe disease of autonomous nervous system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
HF components | 2 hours
  High frequency (HF) components of heartrate-variability in ms²

SECONDARY OUTCOMES:
SDNN | 2 hours
  Standard deviation of normal to normal (SDNN) of heartrate-variability in ms
HF-LF-ratio | 2 hours
  high frequency (HF) to low frequency (LF) ratio of heartrate-variability in 1/s
Tidal volumes | 2 hours
  Changes in mean applicated tidal volumes in ml

OTHER OUTCOMES:
pH | At minute 5, 55, 65 and 115 of the measurement
  pH derived from arterial blood gas analysis
PaO2 | At minute 5, 55, 65 and 115 of the measurement
  Partial pressure of oxygen in mmHg derived from arterial blood gas analysis
PaCO2 | At minute 5, 55, 65 and 115 of the measurement
  Partial pressure of carbon dioxide in mmHg derived from arterial blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Maximlian Schnetzinger, BSc, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT03360968/SAP_000.pdf
  • Study Protocol (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT03360968/Prot_001.pdf